CLINICAL TRIAL: NCT02547116
Title: Epidemiology and Treatment of Small-colony Variant Staphylococcus Aureus in Cystic Fibrosis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Administrative delay
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00047491
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2020-01

CONDITIONS: Cystic Fibrosis; MRSA
MeSH Terms: conditions — Cystic Fibrosis | interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard anti-staphylococcal antibiotic (No Intervention)
- Standard anti-staphylococcal antibiotic + Rifampin (Experimental): Individuals with known, persistent small-colony variant MRSA, who are treated with standard anti-staphylococcal antibiotics, will be treated with their standard therapy in addition to Rifampin.
  Interventions: Drug: Rifampin

INTERVENTIONS:
Drug: Rifampin — Addition of Rifampin to standard anti-Staphylococcal treatment regimen
  Arms: Standard anti-staphylococcal antibiotic + Rifampin

SUMMARY:
Methicillin-susceptible (MSSA) and Methicillin-resistant (MRSA) Staphylococcus aureus (SA) are two of the most important infectious pathogens in CF, with 69% of CF patients having lung infection with MSSA or MRSA in the last year. Wolter and co-workers recently demonstrated that a specific morphologic subtype of MSSA and MRSA, small-colony variant Staph aureus (SCV-SA), is associated with greater decline in lung function and worse clinical outcomes. SCV-SA is already recognized for its ability to contribute to persistent infection, likely due to SCV-SA's ability for intracellular growth, as well as its increased antibiotic resistance compared to normal-colony SA. To investigate the epidemiology and clinical significance of SCV-SA in CF, and explore the hypothesis that SCV-SA may require unique antibiotic treatment strategies to optimize clinical response, the investigators will perform the following:

1. Characterize the epidemiology of SCV-SA infection in both an adult and pediatric CF population and investigate the clinical significance of SCV-SA infection in CF by comparing clinical characteristics and outcomes of CF patients with SCV-SA compared to those with to normal-colony MSSA/MRSA.
2. Characterize the unique microbiologic characteristics of SCV-SA infection in CF by evaluating antibiotic susceptibility profiles and molecular characteristics of SCV-SA in a two large CF patient populations.
3. Perform a 16-patient pilot study of a novel treatment for SCV-SA infection in CF, utilizing low dose rifampin in combination with standard anti-SA antibiotics.

These investigations will delineate the role of SCV-SA as a pathogen in CF and provide guidance to optimize treatment strategies of MSSA/MRSA CF lung infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 12 years of age
2. Confirmed diagnosis of CF based on the following criteria:

   * positive sweat chloride > 60 mEq/liter (by pilocarpine iontophoresis) and/or
   * a genotype with two identifiable mutations consistent with CF or abnormal NPD, and
   * one or more clinical features consistent with the CF phenotype.
3. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
4. Two positive SCV-SA respiratory cultures in the last two years at least six months apart, plus a positive SCV-SA respiratory culture at Screening Visit and Run-in (Day -14) Visit.
5. FEV1 >30% of predicted normal for age, gender, and height at Screening.
6. Weight > 35 kg
7. Females of childbearing potential must agree to practice one highly effective method of birth control, including abstinence. Note: highly effective methods of birth control are those, alone or in combination, that result in a failure rate less than 1% per year when used consistently and correctly. Female patients who utilize hormonal contraceptives as a birth control method must have used the same method for at least 3 months before study dosing. If the patient is using a hormonal form of contraception, patients will be required to also use barrier contraceptives as rifampin can affect the reliability of hormone therapy. Barrier contraceptives such as male condom or diaphragm are acceptable if used in combination with spermicides.

Exclusion Criteria:

1. An acute upper or lower respiratory infection, pulmonary exacerbation, or change in routine therapy (including antibiotics) for pulmonary disease within 14 days of the screening visit.
2. Use of oral or inhaled anti-MRSA drugs within two weeks of the Screening Visit.
3. History of intolerance to rifampin or TMP/SMX, minocycline, and doxycycline.
4. Resistance to rifampin or TMP/SMX, minocycline and doxycycline at screening.
5. Abnormal renal function, defined as creatinine clearance <50 mL/min using the Cockcroft-Gault equation for adults or Schwartz equation in children, at Screening.
6. Abnormal liver function, defined as ≥3x upper limit of normal (ULN), of serum aspartate transaminase (AST) or serum alanine transaminase (ALT), or known cirrhosis. at the time of Screening.
7. Serum hematology or chemistry results which in the judgment of the investigator would interfere with completion of the study.
8. History of or listed for solid organ or hematological transplantation
9. History of sputum culture with non-tuberculous Mycobacteria in the last 6 months.
10. History of sputum culture with Burkholderia Cepacia in the last year.
11. Planned continuous use of soft contact lenses while taking rifampin and no access to glasses.
12. Taking voriconazole and unable to discontinue its use while enrolled in the study.
13. Administration of any investigational drug or device within 28 days of screening or within 6 half-lives of the investigational drug (whichever is longer)
14. Female patients of childbearing potential who are pregnant or lactating, or plan on becoming pregnant
15. Any serious or active medical or psychiatric illness, which in the opinion of the investigator, would interfere with patient treatment, assessment, or adherence to the protocol.
16. Patients taking certain drugs will be excluded from the study:

    a. Drugs, which are contraindicated when rifampin is used (in addition to voriconazole): i. Antiretrovirals: fosamprenavir, atazanavir, lopinavir, saquinavir, nelfinavir, tipranavir, darunavir, rilpivirine,telaprevir, boceprevir, elvitegravir, maraviroc ii. Drugs used to increase systemic exposure of antiretrovirals: Cobicistat iii. Anthelmintic/Antimalarial agents: praziquantel, artemether iv. Antianginal agent: ranolazine v. Psychiatric medications: lurasidone b. Other drugs, not contraindicated, but listed as having major drug to drug interactions i. Antiretrovirals: ritonavir, indinavir, efavirenz, nevirapine, etavirine

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
change in small colony variant Staph. aureus colony forming units on induced sputum respiratory culture | Culture specimens obtained at: Baseline, within 2 weeks of end of standard antibiotic course (control), 1 week prior to intervention, and within 2 weeks of end of intervention

SECONDARY OUTCOMES:
change in lung function, as measured by forced expiratory volume in one second (FEV1) | FEV1 measured at: Baseline, within 2 weeks of end of standard antibiotic course (control), 1 week prior to intervention, and within 2 weeks of end of intervention
patient reported symptoms/quality of life, as captured in the Cystic Fibrosis Questionnaire-Revised (CFQ-R) | CFQ-R administered at: Baseline, within 2 weeks of end of standard antibiotic course (control), 1 week prior to intervention, and within 2 weeks of end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Jennings, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States